CLINICAL TRIAL: NCT01679288
Title: Feasibility of Hand-Held-Ultrasonography in Primary Care in the Screening of Abdominal Aortic Aneurysm and Abdominal Aortic Atheromatosis.
Brief Title: Screening for Abdominal Aortic Aneurysm and Abdominal Aortic Atherosclerosis by Hand-Held Ultrasonography
Acronym: ECO-AAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci d'Atenció Primària de Salut de l'Eixample (Other)
Responsible Party: Principal Investigator, Dr. Antoni Siso Almirall, MD PhD, Consorci d'Atenció Primària de Salut de l'Eixample
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ECO-AAA; ECO-AAA-CAPSE (Registry Identifier: ECO-AAA-CAPSE)
Record Dates: First submitted 2012-06-26; First posted 2012-09-06 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension; Abdominal Aortic Aneurysm; Atheromatosis
Keywords: Hand-Held ultrasonography; Abdominal Aortic Aneurysm; Abdominal Aortic Atherosclerosis; Cardiovascular risk; Primary Health Care
MeSH Terms: conditions — Hypertension; Aortic Aneurysm, Abdominal; Atherosclerosis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ultrasound arm (Experimental): Standardized measurements were made and aorta was tried to be visualized in its entirety, and a minimum of three hard copy images were obtained: upper transverse subxiphoid section, lower transverse section for distal view of aorta, and longitudinal section (with origin of celiac trunk or superior mesenteric artery), determining the maximum diameter in centimeters (cm).
  Interventions: Device: Ultrasound (Trademark:VScan; Manufacturer:General Electrics)

INTERVENTIONS:
Device: Ultrasound (Trademark:VScan; Manufacturer:General Electrics) — Standardized measurements were made and aorta was tried to be visualized in its entirety, and a minimum of three hard copy images were obtained: upper transverse subxiphoid section, lower transverse section for distal view of aorta, and longitudinal section (with origin of celiac trunk or superior mesenteric artery), determining the maximum diameter in centimeters (cm).

SUMMARY:
The purpose of this study is to determine the prevalence of abdominal aortic aneurysm (AAA) and abdominal aortic atheromatosis (AA-At) using a hand-held ultrasound by a general practitioner in Primary Health Care.

DETAILED DESCRIPTION:
Pilot study that prospectively study a cohort of men over 50 years with cardiovascular risk factors: active smokers, former smokers, or hypertensive patients, attended in primary health care center. General Practitioner complete an ultrasonography training in an Ultrasound Unit under supervision of experienced radiologists using an standard ultrasound equipment and hand-held ultrasound (Trademark: VScan®, Manufacturer: General Electric, USA). All images and video recorded are blindly evaluated by a radiologist in order to establish the concordance in the interpretation of images between general practitioner and radiologist. Kappa index is calculated to study the agreement on the presence or absence of AAA and AA-At. Logistic regression analysis is used to determine the factors that influence the presence of AA-At

ELIGIBILITY:
Inclusion Criteria:

* Smokers
* Former smokers.
* Hypertensive patients

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with abdominal aortic aneurysm detected by a Hand-held ultrasound in Primary Care. | 24 months

SECONDARY OUTCOMES:
Number of patients with abdominal aortic atheromatosis detected by Hand-held ultrasound in Primary Care | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Sisó Almirall, MD PhD, Principal Investigator — Consorci d'Atenció Primària de Salut de l'Eixample
Locations (1):
- CAPSE, Barcelona, Barcelona, Spain

REFERENCES:
- See also: Research group's website — http://www.idibaps.org/research/7001/transverse-group-for-research-in-primary-care